CLINICAL TRIAL: NCT01666782
Title: A Randomized Pilot Study Comparing High-Dose Influenza Vaccine to Standard-Dose Influenza Vaccine in Adult Oncology Patients Less Than 65 Years Receiving Chemotherapy
Brief Title: Study Comparing High-Dose Flu Vaccine to Standard Vaccine in Cancer Patients Less Than 65 Receiving Chemotherapy
Acronym: IMMUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saad Jamshed MD (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Saad Jamshed MD, Principal Investigator, Rochester General Hospital
Organization: Rochester General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIC 1336-B12-1
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Influenza Viral Infections
Keywords: Influenza vaccine; Oncology; Chemotherapy
MeSH Terms: conditions — Neoplasms; Influenza, Human | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Dose Influenza Vaccine (Experimental)
  Interventions: Biological: High-Dose Influenza Vaccine
- Standard Trivalent Influenza Vaccine (Active Comparator)
  Interventions: Biological: Standard Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Standard Trivalent Influenza Vaccine — Each 0.5 mL dose contains influenza split virus antigens formulated to contain a total of 45 mcg of influenza virus hemagglutinin, 15 mcg each from the 3 influenza virus strains in the vaccine.One dose given per patient.
  Other Names: Fluzone
  Arms: Standard Trivalent Influenza Vaccine
Biological: High-Dose Influenza Vaccine — Each 0.5 mL dose of Fluzone High-Dose contains influenza split virus antigens that are formulated to contain a total of 180 mcg of influenza virus hemagglutinin, 60 mcg each from the 3 influenza virus strains in the vaccine. One dose given per patient.
  Other Names: Fluzone High-Dose
  Arms: High-Dose Influenza Vaccine

SUMMARY:
The safety and immunogenicity of high dose influenza vaccine has not been studied in young patients receiving chemotherapy. This study will evaluate and compare the immunogenicity and safety of high dose influenza to standard dose influenza vaccine in adult oncology patients who are younger than 65 years old receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old to less than 65 years old
2. Subjects with malignancy must be receiving chemotherapy
3. Medically stable
4. Able to understand and willingness to sign a written informed consent
5. Able to comply with study procedures
6. Life expectancy of more than 3 months
7. Adequate organ function:

   * ANC >1000/mm3
   * Platelet >100,000/uL
   * Creatinine <2 mg/dL
   * AST and ALT <3 times the ULN

Exclusion Criteria:

1. Allergy to eggs
2. Prior allergy to Influenza Vaccine
3. History of Guillain-Barre Syndrome
4. Current febrile illness
5. Other immunosuppressive disease (recipients of solid organ transplant, uncontrolled HIV)
6. Autologous or Allogenic Stem Cell Transplant with in a year
7. Current immunotherapy or immunochemotherapy in the last 6 months (rituximab or ofatumumab)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Jamshed, MD, Principal Investigator — Rochester General Hospital
Locations (2):
- United States (2):
  - Rochester General Hospital, Rochester, New York
  - Lipson Cancer Center Linden Oaks Medical Campus, Rochester, New York

REFERENCES:
- [Derived] Jamshed S, Walsh EE, Dimitroff LJ, Santelli JS, Falsey AR. Improved immunogenicity of high-dose influenza vaccine compared to standard-dose influenza vaccine in adult oncology patients younger than 65 years receiving chemotherapy: A pilot randomized clinical trial. Vaccine. 2016 Jan 27;34(5):630-635. doi: 10.1016/j.vaccine.2015.12.037. Epub 2015 Dec 22. PMID 26721330

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 patients were enrolled but only 100 had evaluable data. 4 patients received a vaccination both in years 1 and 2 of the study- only year 1 results were included in the analysis. 1 additional patient was excluded from the efficacy analysis when it was revealed he had received a second vaccination in the same season.
Period: Overall Study
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Started | 54 | 51
Completed | 50 | 50
Not Completed | 4 | 1
Not completed — Received 2 doses of vaccine | 0 | 1
Not completed — Enrolled both years; year 1 data used | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.94 (7.16) | 52.9 (7.95) | 53.4 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 19 | 24 | 43
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean Titer (GMT) of High-dose Influenza Vaccine vs the Standard Trivalent Influenza Vaccine in Adult Subjects on Chemotherapy Who Are Less Than 65 Years Old.
Description: Measure Hemagglutination Inhibition (HAI) Geometric Mean Titer (GMT) immunogenicity of high-dose (HD) and standard dose (SD) vaccine before and after vaccination at day 28.
Time Frame: Baseline and 28 days
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
titers
  Pre Vaccination H1N1 Antigen | 125.2 [74.6 to 175.8] | 266.1 [52.1 to 480.1]
  Pre Vaccination H3N2 Antigen | 134.1 [54.9 to 213.2] | 143.2 [64.5 to 221.9]
  Pre Vaccination B Antigen | 31.4 [20.4 to 42.3] | 54.7 [31.6 to 77.8]
  Post Vaccination H1N1 Antigen | 1350.1 [819.8 to 1880.4] | 979.1 [609.1 to 1349.0]
  Post Vaccination H3N2 Antigen | 1143.4 [739.6 to 1547.3] | 811.2 [401.2 to 1221.3]
  Post Vaccination B Antigen | 351.6 [215.6 to 487.7] | 228 [129.9 to 326.2]

2. Secondary Outcome: The Seroprotection Rate of High-dose Influenza Vaccine vs Standard Trivalent Influenza Vaccine in Adult Subjects on Chemotherapy Less Than 65 Years Old.
Description: Seroprotection rate was defined as the percentage of patients with a HAI GMT of at least 1:40 28 days after vaccination.
Time Frame: 28 days
Measure: Number; unit: percentage of participants
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
percentage of participants
  H1N1 Antigen | 96 | 90
  H3N2 Antigen | 96 | 96
  B Antigen | 88 | 72

3. Secondary Outcome: The Seroconversion Rate of High-dose Influenza Vaccine Versus Standard Trivalent Influenza Vaccine in Adult Subjects on Chemotherapy Less Than 65 Years Old.
Description: Seroconversion rate was defined as the percentage of patients with a greater than or equal to 4-fold increase in HAI titer 28 days after vaccination.
Time Frame: Baseline and 28 days
Measure: Number; unit: percentage of participants
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
percentage of participants
  H1N1 Antigen | 72 | 46
  H3N2 Antigen | 80 | 58
  B Antigen | 80 | 44

4. Secondary Outcome: Evaluate and Compare the Local Solicited Adverse Events to Both Vaccines.
Description: Local solicited adverse events, standard-dose (SD) vaccine and high-dose (HD) vaccine
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
participants
  Injection site pain- mild | 13 | 10
  Injection site pain-moderate | 3 | 1
  Injection site swelling-mild | 4 | 2
  Injection site swelling-moderate | 1 | 0
  Injection site redness-mild | 2 | 2
  Injection site redness-moderate | 1 | 0
  Injection site itching-mild | 4 | 0
  Injection site itching-moderate | 0 | 0

5. Secondary Outcome: Evaluate and Compare the Systemic Solicited Adverse Events to Both Vaccines.
Description: Systemic solicited adverse events, standard-dose (SD) vaccine and high-dose (HD) vaccine
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
participants
  Fever-mild | 2 | 1
  Fever-moderate | 1 | 1
  Fever-severe | 0 | 0
  Headache-mild | 9 | 12
  Headache-moderate | 6 | 4
  Headache-severe | 1 | 0
  Malaise-mild | 10 | 13
  Malaise-moderate | 10 | 6
  Malaise-severe | 6 | 3
  Myalgia-mild | 12 | 12
  Myalgia-moderate | 8 | 3
  Myalgia-severe | 2 | 1

6. Secondary Outcome: Evaluate and Compare the Local and Systemic Unsolicited Adverse Events to Both Vaccines.
Description: Unsolicited adverse events occurring in more than one patient, standard-dose (SD) vaccine and high-dose (HD) vaccine
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Number analyzed (Participants) | 50 | 50
participants
  Fatigue: Grade 1 or 2 | 6 | 4
  Fatigue: Grade 3 | 1 | 0
  Nausea: Grade 1 or 2 | 3 | 11
  Nausea: Grade 3 | 1 | 0
  Vomiting: Grade 1 or 2 | 2 | 3
  Vomiting: Grade 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: 28 +/- 7 days post-vaccination
Arm/Group | High-Dose Influenza Vaccine | Standard Trivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 26/50 | 22/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Influenza Vaccine (N=50) | Standard Trivalent Influenza Vaccine (N=50)
Malaise (General disorders) | 26 (26) | 22 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 16 (16)
Headache (Nervous system disorders) | 16 (16) | 16 (16)
Injection-site pain (General disorders) | 16 (16) | 11 (11)
Injection-site swelling (General disorders) | 5 (5) | 2 (2)
Injection-site itching (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2)
Injection-site redness (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 11 (11)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All research data and results generated during the course of or as a result of the Research Project shall be the property of Investigator and/or institution. Sanofi Pasteur will have access to the full set of data collected during the Research Project. The text of any manuscript, abstract or oral presentation based on this Research Project will be provided to Sanofi Pasteur at least 30 days prior to submission to a journal, a congress, or prior to an oral presentation.